CLINICAL TRIAL: NCT05802212
Title: Effect of Metformin Intervention on Patients With Polycystic Ovary Syndrome
Brief Title: Effect of Metformin on Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M2021385; 82288102 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2023-02-06; First posted 2023-04-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2023-01

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Volunteers with polycystic ovary syndrome without insulin resistance and intervened with metformin for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin intervention for 12 weeks (Experimental): Metformin intervention for 12 weeks
  Interventions: Drug: Metformin intervention for 12 weeks

INTERVENTIONS:
Drug: Metformin intervention for 12 weeks — PCOS patients were treated with metformin orally for 12 weeks, and various indicators related to fertility were observed.
  Other Names: PCOS patients were treated with metformin for 12 weeks

SUMMARY:
The purpose of the study is to understand the effect of Metformin on patients with PCOS.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of Metformin on reproductive endocrine and reproductive outcomes in women with PCOS, and to explore its underlying mechanisms to provide the intervention strategies for PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are 20 to 40 years old, planning to become pregnant or infertile women.
2. Individuals who are diagnosed as PCOS according to the revised 2003 Rotterdam diagnostic criteria: if 2 out of 3 criteria are met: 1) Oligo- and/or anovulation; 2) Clinical and/or biochemical signs of hyperandrogenism; 3) Polycystic ovaries, and exclusion of other aetiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome).
3. Individuals who can insist on continuous monitoring in the outpatient clinic. Individuals who are not participating in other research projects currently or 3 months before the intervention.
4. Volunteers with polycystic ovary syndrome without insulin resistance.

Exclusion Criteria:

1. Individuals who suffering from other diseases that may cause hyperandrogenism and ovulation abnormalities.
2. Individuals who are during pregnant, lactation or menopause.
3. Individuals who currently receiving weight-loss drugs or surgery or within the past 2 months.
4. Individuals who take niacin, nicotinamide, or other vitamin B3-related supplementation currently or within the past 2 months.
5. Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
6. Use of medications that affect hormone levels, appetite, carbohydrate absorption, and metabolism within the past 2 months.
7. Individuals with severe liver diseases or kidney disease that are ineligible to participate in the study.
8. A medical history of severe cardiovascular and cerebrovascular diseases.
9. Individuals who currently suffer from severe gastrointestinal diseases or undergo gastrointestinal resection that may affect nutrient absorption.
10. Individuals who drink more than 15g of alcohol per day or have a smoking habit.
11. Individuals who need drug treatment for any mental illness such as epilepsy and depression.
12. Cancer patients.
13. Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Luteinizing hormone in serum | before and after 2, 12 weeks of intervention
  Changes of luteinizing hormone(mIU/mL) in serum after the intervention.
4-Androstenedione in serum | before and after 2, 12 weeks of intervention
  Changes of 4-Androstenedione(pmol/L) in serum after the intervention.

SECONDARY OUTCOMES:
Testosterone in serum | before and after 2, 12 weeks of intervention
  Changes of testosterone(nmol/L) in serum after the intervention.
Estradiol in serum | before and after 2, 12 weeks of intervention
  Changes of estradiol(pmol/L) in serum after the intervention.
Prolactin in serum | before and after 2, 12 weeks of intervention
  Changes of prolactin(ng/mL) in serum after the intervention.
Follicle number | after 12 weeks of intervention
  The number of all antral follicles in each ovary will be determined using transvaginal ultrasonography for each participant.
Follicle number | before intervention
  The number of all antral follicles in each ovary will be determined using transvaginal ultrasonography for each participant.
Ovarian volume | after 12 weeks of intervention
  The size of each ovary will be determined using transvaginal ultrasonography for each participant in early follicular phase.
Ovarian volume | before intervention
  The size of each ovary will be determined using transvaginal ultrasonography for each participant in early follicular phase.
The alterations of plasma lipid metabolites | after 12 weeks of intervention
  Determination the alterations of lipid metabolites before and after metformin intervention by metabolomics.
The alterations of plasma lipid metabolites | after 2 weeks of intervention
  Determination the alterations of lipid metabolites before and after metformin intervention by metabolomics.
The alterations of plasma lipid metabolites | before intervention
  Determination the alterations of lipid metabolites before and after metformin intervention by metabolomics.
Fasting insulin | before and after 2, 12 weeks of intervention
  Changes in plasma insulin concentration after the intervention.
Blood sugar level | before and after 2, 12 weeks of intervention
  Changes in plasma glucose concentration after the intervention.
The alterations of secondary metabolites of gut fungi and bacteria | after 12 weeks of intervention
  Determination the alterations of secondary metabolites of gut fungi and bacteria before and after metformin intervention by metabolomics
The alterations of secondary metabolites of gut fungi and bacteria | after 2 weeks of intervention
  Determination the alterations of secondary metabolites of gut fungi and bacteria before and after metformin intervention by metabolomics
The alterations of secondary metabolites of gut fungi and bacteria | before intervention
  Determination the alterations of secondary metabolites of gut fungi and bacteria before and after metformin intervention by metabolomics
The species and genus abundance changes of fungi and bacteria gut microbiota composition | before and after 2, 12 weeks of intervention
  Determination the species and genus abundance changes of gut microbiota among before and after intervention by ITS genomic
Follicular stimulating hormone in serum | before and after 2, 12 weeks of intervention
  Changes of follicular stimulating hormone(mIU/mL) in serum after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Qiaojie, Professor, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No